CLINICAL TRIAL: NCT03498781
Title: The Impact of Multiple Behavior Change on the Effectiveness of Implementation Intentions to Promote Fitness Center Visitation
Brief Title: Good Intentions Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of interest in pool of potential participants
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: GFHNRC408
Record Dates: First submitted 2018-03-29; First posted 2018-04-17 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Obesity; Overweight
Keywords: Exercise
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study will be a between group factorial design. The between subjects variable will be group assignment. The within subjects variable will be time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise-only intervention (Experimental): Participants will receive information regarding the health benefits of regular aerobic and resistance training exercise and current physical activity guidelines for adults.
  Interventions: Other: Exercise-only
- Control intervention (Sham Comparator): Participants will receive information regarding the health risks of chronic stress as well as suggested methods to reduce stress.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise-only — Participants will write goals related to exercise, the most desired outcome of reaching their goals, anticipated obstacles/barriers which may prevent them from achieving their goals, and if-then statements proactively describing how to overcome or avoid obstacles.
  Arms: Exercise-only intervention
Other: Control — Participants will be asked to identify stress-reduction techniques which they can use in their daily lives and will be encouraged to practice them as necessary.
  Arms: Control intervention

SUMMARY:
The purpose of this study is to explore the effects of an intervention designed to help increase physical activity and decrease screen time.

DETAILED DESCRIPTION:
The purpose of this study is to investigate attendance, exercise, and screen time habits in fitness center members. Because they are the population under investigation, recruitment will take place via the fitness center facilities. This population is under investigation because much of this population is sedentary and does not exercise at recommended levels, despite access to physical fitness facilities. This research will investigate methods to encourage physical activity in this population.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index from 18-45 kg/m2

Exclusion Criteria:

* have any medical conditions that prevent participant from safely taking part in physical activity
* currently a smoker
* are pregnant, breastfeeding, or plan to become pregnant
* have visited fitness centers more than eight times in the past two months
* exercise outside of fitness centers more than once a week for one hour at a time in the past month
* do not engage in more than 14 hours a week of screen-based activities
* do not have a primarily sedentary job

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Fitness center attendance | Week 0, 8, 16
  Change in fitness center attendance as measured by number of visits per week

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No